CLINICAL TRIAL: NCT02893423
Title: The Dose Dependent Effect of Ropivacaine Transversus Abdominis Plane Blocks on Postoperative Analgesia After Cesarean Section
Brief Title: Ropivacaine Transversus Abdominis Plane Blocks for Cesarean Section Analgesia
Acronym: TAPROPI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A better study with a better drug was started and thus this study was terminated
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, kalpana tyagaraj, Residency Program Director, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Study # 13/01/VA01
Record Dates: First submitted 2016-06-26; First posted 2016-09-08 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Pain
Keywords: Ropivacaine; C-Section Analgesia; Tap Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 - 0.5% Ropivacaine (Active Comparator): Patients will receive 0.5% Ropivacaine for the TAP block Procedure: Ultrasound guided TAP BLOCK Drug: 0.5% ropivacaine 20ml of 0.5% ropivacaine is used to perform the TAP block Other Names: •Naropin
  Interventions: Drug: Ropivacaine
- Group 2 - 0.25% Ropivacaine (Active Comparator): Patients will receive 0.25% for the TAP block Procedure: ULTRASOUND GUIDED TAP BLOCK Drug: 0.25% ropivacaine 20ml of 0.25% ropivacaine is used to perform the TAP block Other Names: •Naropin
  Interventions: Drug: Ropivacaine
- Group 3 - No Tap Block (No Intervention): Patients will not receive a TAP BLOCK

INTERVENTIONS:
Drug: Ropivacaine — Using 2 Different Concentrations of Ropivacaine in Tap Block for Postoperative Analgesia for C-Section Patients
  Other Names: Naropin
  Arms: Group 1 - 0.5% Ropivacaine; Group 2 - 0.25% Ropivacaine

SUMMARY:
With this research the investigators hope to determine the lowest dose of ropivacaine used in transversus abdominis plane (TAP) blocks that can effectively treat pain in women after cesarean section (c-section).

DETAILED DESCRIPTION:
With this research the investigators hope to determine the lowest dose of ropivacaine used in transversus abdominis plane (TAP) blocks that can effectively treat pain in women after cesarean section (c-section). The TAP is a space between the muscle layers of the abdominal wall that houses nerves supplying the abdominal skin. The investigators will inject the local anesthetic ropivacaine into this space to freeze these nerves and prevent pain following c-section. The investigators will compare three different doses of ropivacaine (0.5%, 0.25%, 0%) to determine the lowest dose that controls pain with the fewest side effects. Participants in this study will receive 0.5% (Group 1), 0.25% (Group 2), or 0% (Group 3) ropivacaine TAP blocks to control pain after c-section. At 2, 6, 12, 24, and 48 hours after cesarean section visual analog pain scores (VAS) for pain on movement, pain at rest, and pain with cough will be collected along with the time to first postoperative analgesic request, patient satisfaction scores, and patient demographics. The analgesic regimen will be considered effective if it provides lower average visual analog scores for pain with movement. Secondary outcomes will be higher patient satisfaction, better pain control, fewer postoperative analgesic requests, and fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients undergoing elective c-section

Exclusion criteria:

* Allergy to local anesthetics
* Contraindication to tap blocks

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KALPANA TYAGARAJ, MD, Principal Investigator — MAIMONIDES MEDICAL CENTER, 4802, 10TH AVENUE, BROOKLYN, NY-11219
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - 0.5% Ropivacaine | Group 2 - 0.25% Ropivacaine | Group 3 - No Tap Block
Started | 17 | 16 | 18
Completed | 17 | 16 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - 0.5% Ropivacaine | Group 2 - 0.25% Ropivacaine | Group 3 - No Tap Block | Total
Number analyzed (Participants) | 17 | 16 | 18 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.65 (6.30) | 29.17 (4.29) | 31.0 (4.72) | 30.94 (5.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 18 | 51
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 18 | 51

OUTCOME MEASURES:

1. Primary Outcome: POSTOPERATIVE PAIN
Description: Severity of postoperative pain will be assessed using(VAS) scale. Post-operative pain scale name: Visual Analog Scale (0-10) with 0 being no-pain and 10 being maximum pain.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 - 0.5% Ropivacaine | Group 2 - 0.25% Ropivacaine | Group 3 - No Tap Block
Number analyzed (Participants) | 17 | 16 | 18
score on a scale | 2.35 (3.08) | 1.94 (2.77) | 0.56 (.922)

ADVERSE EVENTS:
Arm/Group | Group 1 - 0.5% Ropivacaine | Group 2 - 0.25% Ropivacaine | Group 3 - No Tap Block
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No